CLINICAL TRIAL: NCT06744686
Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of HT-102Injection in Healthy Subjects and Hepatitis B E Antigen-Negative Patients with Chronic Hepatitis B Virus Infection: a Randomized, Double-blind, Placebo-controlled, Single and Multiple Subcutaneous Injections, and Dose Escalation Phase 1 Clinical Study
Brief Title: Phase 1 Study of HT-102 Administered Subcustaneously in Healthy Participants and Patients with Chronic Hepatitis B for Safety, Tolerability, Pharmacokinetics (PK), and Antiviral Activity (only in Participants with Chronic HBV Infection)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou HepaThera Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT-102-101
Record Dates: First submitted 2024-12-09; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A (Healthy participants administered with HT-102 or placebo) (Experimental): Healthy participants in all dose groups were randomly assigned to receive a single dose of HT-102 or placebo subcutaneously
  Interventions: Drug: HT-102; Drug: Placebo
- Part B (Patients with CHB administered with HT-102 or placebo) (Experimental): Patients with chronic hepatitis B in all dose groups were randomly assigned to receive 5 dose of HT-102 or placebo subcutaneously every week.
  Interventions: Drug: HT-102; Drug: Placebo

INTERVENTIONS:
Drug: HT-102 — 50mg, 150mg, 300mg, 600mg
  Arms: Part A (Healthy participants administered with HT-102 or placebo)
Drug: HT-102 — 50mg, 150mg, 300mg
  Arms: Part B (Patients with CHB administered with HT-102 or placebo)
Drug: Placebo — Placebo

SUMMARY:
Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of HT-102 (BM012) Injection in Healthy Subjects and Hepatitis B e Antigen-Negative Patients with Chronic Hepatitis B Virus Infection: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Subcutaneous Injections, and Dose Escalation Phase 1 Clinical Study

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants SAD:

* Male participants weighed ≥ 50.0 kg, female participants weighed ≥ 45.0 kg;
* Participants were healthy individuals;
* Participants promise to have no plans to have a child, donate sperm or eggs and voluntarily take effective non-drug contraception measures during the trial and within 3 months after the end of the trial;

Participants with Chronic HBV infection, MAD:

* Chronic HBV infection, and HBeAg negative;
* Patients who had received antiviral therapy for at least one year before screening and stabilization therapy with nucleoside (nucleotide) reverse transcriptase inhibitors for ≥ 3 months before screening (nucleoside (nucleotide) reverse transcriptase inhibitors;

Exclusion Criteria:

* Participants with a history of active pathological hemorrhage or those with bleeding tendency, or those with a history of neurological disease;
* Participants with major trauma or major surgery within 3 months before trial screening;
* Participants with a history of drug allergy;
* Participants who used any drugs before trial screening or are using any drugs, including vitamins and Chinese herbal medicines;
* Participants with abnormal results of ECG examination, laboratory test in the screening period which were judged as clinically significant;
* Participants who cannot tolerate subcutaneous injection;
* Patients with a previous clinical diagnosis of liver cirrhosis, or a history of alcoholic liver disease, autoimmune liver disease, inherited metabolic liver disease, and other liver diseases;
* Participants with a clinically significant acute infection;
* Women who were pregnant or lactating or had a positive pregnancy test result;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From administration to the end of treatment at 8 weeks
Time to Reach Maximum Plasma Concentration (Tmax) | From administration to the end of treatment at 8 weeks

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | From administration to the end of treatment o at 10 weeks
Area Under the Plasma Concentration Versus Time Curve (AUC) | From administration to the end of treatment o at 10 weeks
Apparent Terminal Elimination Half-life (T1/2) | From administration to the end of treatment o at 10 weeks
Apparent Plasma Clearance (CL/F) | From administration to the end of treatment o at 10 weeks
Apparent volume of distribution（Vd/F） | From administration to the end of treatment o at 10 weeks
Change of Serum HBsAg From Baseline | From administration to the end of treatment o at 10 weeks
Change of Serum HBV DNA From Baseline | From administration to the end of treatment o at 10 weeks
Change of Serum HBV RNA From Baseline | From administration to the end of treatment o at 10 weeks
Change of Serum HBcrAg From Baseline | From administration to the end of treatment o at 10 weeks
Change of Serum HBcAb From Baseline | From administration to the end of treatment o at 10 weeks
Titers of Anti-drug Antibody (ADA) to HT-102 | From administration to the end of treatment o at 10 weeks
  ADA analysis for predose and 8week (Part A) or 10weeks (Part B) postdose

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - People's Hospital of Qingyuan, Qingyuan, Guangdong
  - Luoyang Central Hospital, Luoyang, Henan
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No